CLINICAL TRIAL: NCT04916041
Title: Visual Function in Subjects Implanted With Advanced Technology Intraocular Lenses
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clínica Rementería (Other)
Responsible Party: Sponsor
Other Study IDs: 21/365-O_P
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Lenses, Intraocular
MeSH Terms: interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (5):
- Vivity: Patients who have undergone bilateral implantation of Vivity intraocular lens
  Interventions: Device: Cataract surgery with bilateral implantation of the same type of intraocular lens
- Eyhance: Patients who have received bilateral implantation of an Eyhance intraocular lens
  Interventions: Device: Cataract surgery with bilateral implantation of the same type of intraocular lens
- EMV: Patients who have undergone bilateral implantation of Vivity intraocular lens
  Interventions: Device: Cataract surgery with bilateral implantation of the same type of intraocular lens
- Panoptix: Patients who have undergone bilateral implantation of Panoptix intraocular lens
  Interventions: Device: Cataract surgery with bilateral implantation of the same type of intraocular lens
- Rayner Trifocal: Patients who have undergone bilateral implantation of Rayner trifocal intraocular lens
  Interventions: Device: Cataract surgery with bilateral implantation of the same type of intraocular lens

INTERVENTIONS:
Device: Cataract surgery with bilateral implantation of the same type of intraocular lens — Cataract surgery with bilateral implantation of the same type of intraocular lens

SUMMARY:
Multiple intraocular lens are nowadays available for implantation after cataract surgery. They use different technology to try to improve patient spectacle independence. It is necessary to better characterise the performence of each type of lens, as well as to define how they are affected by residual refractive errors. The purpose of this study is to evaluate visual function in patients implanted with different lenses (advanced monofocals, trifocals) in order to be able to recommend the best type of lens for each patient.

ELIGIBILITY:
Inclusion Criteria: Bilateral cataract surgery Bilateral implantation of one of the intraocular lens models included in the study

Exclusion Criteria:

Intrasurgical complications Postsurgical complications Ophthalmological disease that limits visual potential as estimated by investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone bilateral cataract surgery between three and nine months prior to study procedures, with bilateral implantation of one of the intraocular lens models included in the study
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Intermediate binocular uncorrected visual acuity | 3-9 months after cataract surgery

SECONDARY OUTCOMES:
Distance binocular uncorrected visual acuity | 3-9 months after cataract surgery
Near binocular uncorrected visual acuity | 3-9 months after cataract surgery
Binocular contrast sensitivity | 3-9 months after cataract surgery
Halo perception | 3-9 months after cataract surgery
Self-reported visual function questionnaires | 3-9 months after cataract surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Rementería, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No